CLINICAL TRIAL: NCT01056926
Title: Neurobiology of Nicotine and Non-nicotine Components of Tobacco Addiction
Acronym: NNN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00004092
Record Dates: First submitted 2010-01-14; First posted 2010-01-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2013-07

CONDITIONS: Smoking
Keywords: smoking; nicotine; Effects of nicotine and non-nicotine factors on continuous working memory.; Effects of nicotine and non-nicotine factors on cue reactivity.; Use of nicotine patches, placebo patches, and denicotinized cigarettes.; memory
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine Patch + Denic Smoking (Experimental): Subjects will wear a nicotine patch and smoke denic cigarettes for 24 hours prior to scan
  Interventions: Drug: Nicotine patch
- Placebo Patch + Denic Smoking (Experimental): Subjects will wear a placebo patch and smoke denic cigarettes 24 hours prior to scan
  Interventions: Drug: Placebo Patch
- Nicotine Patch + No Smoking (Experimental): Subjects will wear a nicotine patch and not smoke for 24 hours prior to scan
  Interventions: Behavioral: Quit smoking; Drug: Nicotine patch
- Placebo Patch + No Smoking (Experimental): Subjects will wear a placebo patch and not smoke for 24 hours prior to scan
  Interventions: Behavioral: Quit smoking; Drug: Placebo Patch

INTERVENTIONS:
Behavioral: Quit smoking — Subjects will quit smoking for 2 fMRIs, each abstinence lasting 2 days
  Arms: Nicotine Patch + No Smoking; Placebo Patch + No Smoking
Drug: Nicotine patch — Subjects will wear a 21mg patch for 2 fMRIs, each condition lasting 2 days. They will take the patch off at night.
  Arms: Nicotine Patch + Denic Smoking; Nicotine Patch + No Smoking
Drug: Placebo Patch — Subjects will wear a placebo patch for 2 fMRIs, each condition lasting 2 days. They will take the patch off at night.
  Arms: Placebo Patch + Denic Smoking; Placebo Patch + No Smoking

SUMMARY:
In the present study the investigators will measure the effects of nicotine and non-nicotine factors on brain function during cognitive processes that are differentially sensitive to these factors. One process-continuous working memory (CWM)-is implemented via a network of frontal and parietal brain regions and is highly dopamine dependent. Smoking cessation results in significant deficits in CWM which can persist for weeks and are reversed by resumption of nicotine administration in the form of smoking or nicotine replacement. Additionally, CWM deficits are observed during smoking of denic cigarettes. Brain function during CWM is modulated by smoking abstinence and subsequent nicotine administration and activity in the dlPFC is implicated in these effects. Collectively, these data suggest that CWM is highly sensitive to the nicotine, but not non-nicotine components of smoking. Brain function during CWM is altered by smoking abstinence and nicotine, but the effect of smoking, in the absence of nicotine, has not been evaluated.

Another process-cue-reactivity (CR)-results from the repeated pairing of otherwise neutral stimuli with nicotine administration. Acute smoking cessation has not been shown to have strong effects on CR in the form of cue-provoked craving, nor has nicotine replacement been shown to have robust effects on CR. Likewise, the direct effects of smoking abstinence on brain CR have been small; though craving has been shown to modulate relations between abstinence and CR. Moreover, recent data from our lab suggest larger 'doses' of abstinence (~ 24 hrs) may amplify brain responses to cues. The effect of smoking in the absence of nicotine, on CR has not, to our knowledge, been evaluated. Collectively, these data suggest that CR in the form of cue-induced craving is not highly sensitive to the effects of short-term smoking abstinence or nicotine. Brain CR is modulated by abstinence-induced craving and longer-term abstinence, but it is unclear whether abstinence from nicotine or non-nicotine components is responsible for these effects.

In the present study, we propose to evaluate the effects of non-nicotine and nicotine factors on CWM and CR using functional magnetic resonance imaging. This method allows for the non-invasive assessment of brain function. We will also examine the role of genes in moderating and mediating the effects of nicotine and non-nicotine factors on cognitive function

DETAILED DESCRIPTION:
Overview. In a fully factorial design, thirty-six (n=36) adult smokers will undergo fMRI scanning at least 24 hours after each of the following conditions: 1) Nicotine Patch + Denic Smoking, 2) Placebo Patch + Denic Smoking, 3) Nicotine Patch + No Smoking, and 4) Placebo Patch+ No Smoking. During scanning, participants will complete a laboratory based measure of continuous working memory (n-back)-a measure of continuous working memory-and the cue-reactivity task (CR)-a measure of responses to smoking cues. Broadly, we hypothesize 1) abstinence from nicotine, regardless of smoking, will disrupt CWM performance and brain function, 2) abstinence from nicotine and denics will potentiate brain CR but differentially contribute to this effect and 3) that individual differences in smoking behavior and motivation will predict the effects of nicotine and non-nicotine factors on brain function.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy,
2. between the ages of 18 and 55,
3. smoking of at least 10 cigarettes/day of a brand delivering > 0.5 mg nicotine according to the standard Federal Trade Commission (FTC) method,
4. an afternoon expired carbon monoxide concentration of at least 10 ppm (to confirm inhalation),
5. no interest in quitting smoking as measured by self-report, and
6. right-handed as measured by a three-item scale used in our laboratory.

Exclusion Criteria:

1. inability to attend all required experimental sessions,
2. significant health problems (e.g., chronic hypertension, emphysema, seizure disorder, history of significant heart problems),
3. use of psychoactive medications,
4. use of smokeless tobacco,
5. current alcohol or drug abuse,
6. use of illegal drugs as measured by urine drug screen,
7. current use of nicotine replacement therapy or other smoking cessation treatment,
8. presence of conditions that would make MRI unsafe (e.g., pacemaker),
9. presence of conditions contraindicated for nicotine replacement therapy (e.g., skin allergies or disorders).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Measure cue reactivity while subjects undergo a functional magnetic resonance imaging (fMRI). | 1.25 hours

SECONDARY OUTCOMES:
Measure continuous working memory while subjects are scanned in a functional magnetic resonance imaging (fMRI). | 1.25 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States